CLINICAL TRIAL: NCT07301931
Title: A Modified Chair Technique for Acute Anterior Shoulder Dislocation Compare With Traction-counter Traction Technique : A Randomized Controlled Trial
Brief Title: A Modified Chair Technique for Acute Anterior Shoulder Dislocation Compare With Traction-counter Traction Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen Hospital (Other Government)
Responsible Party: Principal Investigator, Pawat Yuwamitr, Orthopedic, Khon Kaen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEF66038
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Anterior Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified chair technique (Active Comparator)
  Interventions: Procedure: Modified chair technique
- traction-counter traction teahnique (Active Comparator)
  Interventions: Procedure: Traction-counter traction technique

INTERVENTIONS:
Procedure: Modified chair technique — Modified Chair Technique is a closed reduction method for acute anterior shoulder dislocation that adapts the traditional chair technique to improve convenience and safety in the emergency setting. Instead of using a standard chair backrest, this modified approach utilizes the side rail of a patient transport stretcher, which serves as a stable fulcrum beneath the patient's axilla.
  Arms: Modified chair technique
Procedure: Traction-counter traction technique — Traction-Counter Traction Technique is applying longitudinal traction to the affected arm while simultaneously providing counter traction across the patient's torso, allowing controlled separation of the humeral head from surrounding soft tissues to facilitate reduction.
  Arms: traction-counter traction teahnique

SUMMARY:
Anterior shoulder dislocation is the most common type of joint dislocation and requires timely and effective closed reduction. The traction-counter traction technique is widely used in Thailand, although it may require patient transfer and sedation, which can increase the risk of adverse events. The modified chair technique has been introduced as a simpler, potentially more convenient method that may allow reduction to be performed in a single location

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with anterior shoulder dislocation based on physical examination and radiographic findings, including both first-episode (primary) and recurrent cases.
* Patients aged 18 years or older.
* Patients who are fully conscious and able to provide informed consent.
* Patients with a Glasgow Coma Score (GCS) of 15.

Exclusion Criteria:

* Patients with a history of seizure prior to the current injury.
* Patients with vascular or neurological deficits detected on physical examination.
* Patients with associated humeral fractures identified on radiographic imaging.
* Patients with multiple traumatic injuries involving.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
To compare the success rate of shoulder reduction between the modified chair technique and the traction-counter traction technique in patients with acute anterior shoulder dislocation. | immediate after procedure

SECONDARY OUTCOMES:
To compare the level of pain during the shoulder reduction procedure between the modified chair technique and the traction-counter traction technique. | immediate after procedure
  we record pain with visual analog scale range from 0 to 10
Evaluate the complications associated with shoulder reduction from using the modified chair technique and the traction-counter traction technique. | 30 minute after procedure
  Complication such as brachial plexus injury, proximal humerus fracture, muscle spasm

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen Hospital, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dreu M, Aufmesser W, Aufmesser H, Dolcet C, Feigl G, Sadoghi P. A simple and gentle technique for reduction after anterior shoulder dislocation. Arch Orthop Trauma Surg. 2015 Oct;135(10):1379-84. doi: 10.1007/s00402-015-2279-6. Epub 2015 Jul 21. PMID 26193846
- [Result] Smith SL. An investigation comparing the Oxford Chair Technique with the traditional methods of glenohumeral dislocation reduction currently implemented. Int Emerg Nurs. 2009 Jan;17(1):38-46. doi: 10.1016/j.ienj.2008.09.004. Epub 2008 Nov 25. PMID 19135014
- [Result] Sayegh FE, Kenanidis EI, Papavasiliou KA, Potoupnis ME, Kirkos JM, Kapetanos GA. Reduction of acute anterior dislocations: a prospective randomized study comparing a new technique with the Hippocratic and Kocher methods. J Bone Joint Surg Am. 2009 Dec;91(12):2775-82. doi: 10.2106/JBJS.H.01434. PMID 19952238
- [Result] Mahirogullari M, Akyildiz F, Koksal I, Cakmak S, Kurklu M, Kuskucu M. Chair method: a simple and effective method for reduction of anterior shoulder dislocation. Acta Orthop Traumatol Turc. 2012;46(2):102-6. doi: 10.3944/AOTT.2012.2676. PMID 22491434
- [Result] Ghane MR, Hoseini SH, Javadzadeh HR, Mahmoudi S, Saburi A. Comparison between traction-countertraction and modified scapular manipulation for reduction of shoulder dislocation. Chin J Traumatol. 2014 Apr 1;17(2):93-8. PMID 24698578
- [Result] Guler O, Ekinci S, Akyildiz F, Tirmik U, Cakmak S, Ugras A, Piskin A, Mahirogullari M. Comparison of four different reduction methods for anterior dislocation of the shoulder. J Orthop Surg Res. 2015 May 28;10:80. doi: 10.1186/s13018-015-0226-4. PMID 26016671
- [Result] Fennelly JT, Gourbault L, Neal-Smith G, Pradhan A, Gade V, Baxter JA. A systematic review of pre-hospital shoulder reduction techniques for anterior shoulder dislocation and the effect on patient return to function. Chin J Traumatol. 2020 Oct;23(5):295-301. doi: 10.1016/j.cjtee.2020.08.003. Epub 2020 Aug 12. PMID 32893114
- [Result] Cunningham NJ. Techniques for reduction of anteroinferior shoulder dislocation. Emerg Med Australas. 2005 Oct-Dec;17(5-6):463-71. doi: 10.1111/j.1742-6723.2005.00778.x. PMID 16302939
- [Result] Alkaduhimi H, van der Linde JA, Willigenburg NW, van Deurzen DFP, van den Bekerom MPJ. A systematic comparison of the closed shoulder reduction techniques. Arch Orthop Trauma Surg. 2017 May;137(5):589-599. doi: 10.1007/s00402-017-2648-4. Epub 2017 Mar 1. PMID 28251280